CLINICAL TRIAL: NCT04674423
Title: The Effectiveness and Safety of Tenofovir Alafenamide in the Treatment of Chronic Hepatitis B Patients With Mildly Elevated Alanine Aminotransferase and Significant Liver Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB-CR 108-062
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-07

CONDITIONS: Chronic Hepatitis b
Keywords: Chronic hepatitis B, tenofovir Alafenamide, ALT, liver injury
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Masking Description: Two treatment groups: TAF group and control group
  Treatment groups:
  1. TAF treatment group (144 weeks)
  2. Controlled group (144 weeks)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAF Treatment (Experimental): TAF treatment for 144 weeks and followed for 48 weeks after 144-week TAF treatment
  Interventions: Drug: Tenofovir Alafenamide
- Observation arm (No Intervention): Observation for 144 weeks

INTERVENTIONS:
Drug: Tenofovir Alafenamide — Tenofovir Alafenamide treatment for 144 weeks
  Arms: TAF Treatment

SUMMARY:
In Taiwan, non-cirrhosis CHB patients with mildly elevated ALT are not candidates for antiviral treatment under Taiwan NIH reimbursement criteria. Disease severity could range from mildly liver injury to cirrhosis in this group of patients. There is a substantial population of patients required antiviral treatment, but not fulfill the criteria of reimbursement treatment.

For the 2 phase 3 trials of TAF, the treatment criteria of ALT were more than 2x of ULN and did not included liver biopsy as a pre-treatment assessment. In this study, CHB patient with ALT level of 1-2x ULN and significant liver injury evaluated by liver biopsy is the target study population.

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1. Overview Hepatitis B virus (HBV) infection could lead to chronic hepatitis, liver cirrhosis, and hepatocellular carcinoma (HCC). Liver diseases and its complications remains one of the leading causes of death in Taiwan. Epidemiology study shows that HBV viral load is positively associated with incidence of cirrhosis and HCC in the long-term follow-up. Several lines of evidence also revealed that effective control of HBV could reduce the risk of liver decompensation and HCC. Currently, treatment of chronic hepatitis B (CHB) includes pegylated interferon (IFN) and nucleoside or nucleotide analogues (NUC). NUC treatment exhibits the advantages of easy, safe, wide ranges of indications, and strong viral suppression when compared with IFN.

   1.2. Clinical experience of NUC treatment The first line of NUC treatment currently are entecavir (ETV), tenofovir disoproxil fumarate (TDF), and tenofovir alafenamide (TAF). All these drugs are effective in viral suppression, maintain normal aminotransferase, and exhibit long term safety and minimal viral resistance in treatment for HBeAg positive, HBeAg negative, and cirrhosis patients. Fibrosis improvement and cirrhosis reversion could be achieved in a significant proportion of patients treated with 5-year of ETV or TDF. Some safety concern raised. Renal function deterioration and decreased bone mineral density are present in patient with human immunodeficiency virus (HIV) infection and treated with TDF containing regimen. In CHB patients, impairment of renal function occurs in 1-2% of 8-years TDF treatment. There are controversies in relationship between TDF and bone mineral density. The safety issues of long-term TDF treatment, except its high efficacy in viral suppression, still remains and needs to monitor during treatment course. 1.3. Clinical experience of TAF TAF is a new nucleotide analogue. Two phase III trials, study 108 and 110, were designed to compare the efficacy and safety of TAF and TDF in HBeAg positive and HBeAg negative chronic hepatitis B patients. After two years of treatment, similar viral suppression, but more rapid and higher percentages achieved normalization of alanine aminotransferase (ALT) were observed in TAF group. In addition, renal function measured by estimated glomerular filtration rate (eGFR) was maintained in TAF group. In contrast, TDF group exhibited decline of eGFR. Similarly, bone mineral measured by dual-energy x-ray absorptiometry (DEXA) was maintained TAF group, but decreased in TDF group. In EASL practical guideline for management of chronic hepatitis C suggests that patients with age more than 60 years, bone diseases, and renal alterations should select TAF over TDF.

   1.4. Current treatment criteria for non-cirrhosis CHB In APASL and AASLD treatment guideline for CHB, both suggested that non-cirrhosis patients with significant viral load and ALT >2x upper limit of normal range (ULN) in either HBeAg positive or HBeAg negative should be treated. The significant viral load is defined as HBV DNA >20000 IU/mL in HBeAg positive and HBV DNA >2000 IU/mL in HBeAg negative. Current reimbursement criteria of Taiwan NIH also follow these conditions. For those non-cirrhotic patients with significant HBV viral load and ALT level between 1-2x of ULN, treatment is not reimbursed under the NIH criteria. However, treatment should be commenced by liver histology severity which is defined as significant liver inflammation or fibrosis according to APASL and AASLD guidelines.

   1.5. Rationale of study In Taiwan, non-cirrhosis CHB patients with mildly elevated ALT are not candidates for antiviral treatment under Taiwan NIH reimbursement criteria. Disease severity could range from mildly liver injury to cirrhosis in this group of patients. There is a substantial population of patients required antiviral treatment, but not fulfill the criteria of reimbursement treatment.

   For the 2 phase 3 trials of TAF, the treatment criteria of ALT were more than 2x of ULN and did not included liver biopsy as a pre-treatment assessment. In this study, CHB patient with ALT level of 1-2x ULN and significant liver injury evaluated by liver biopsy is the target study population.
2. STUDY DESIGN 2.1. Study population This is a phase 4, multicenter, open label study at 12 academic hospitals in Taiwan. Treatment naïve CHB patients with mildly elevated ALT (1-2x of ULN) and significant liver injury evaluated by liver biopsy will be enrolled. The study will be approved by Institutional Review Board (IRB) and will be conducted in accordance with the principles of Declaration of Helsinki and the international Conference on Harmonization for Good Clinical Practice. Informed consent will be provided before enrollment for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20 years
* Presence of HBsAg positivity for more than 6 months that indicated chronic HBV infection;
* HBV viral load more than 20000 IU/mL in HBeAg positive or more than 2000 IU/mL in HBeAg Negative CHB patients;
* Presence of liver injury which was defined as histology activity index (HAI) >3 by Knodell necroinflammantion scoring system or liver fibrosis stage 2 or stage 3 by Metavir scoring system; Liver histology available for evaluation 6 months before starting screening is also acceptable. This criteria is limited to subjects enrolling TAF treatment group.
* ALT level between 1-2 folds of ULN for at least one occasion in recent 1 year before screening;
* Treatment naïve;

Exclusion Criteria:

* Other etiology of chronic hepatitis; Those patients with spontaneous clearance of HCV defined as presence of anti-HCV antibody but undetectable of HCV RNA at least 3 months before enrollment and without history of anti-viral treatment could be included.
* Severe comorbid disorders;
* Uncontrolled diabetes mellitus (HBA1c > 8.5%);
* Current evidence or suspicious of malignancy;
* Diagnosis of liver cirrhosis;
* eGFR < or = 30 ml/min/1.73m2.
* Any one of following hematology or biochemical or clinical abnormalities:

Albumin <3.5g/dL, Total Bilirubin >2.5mg/dL, prothrombin time prolongation >4 sec or INR >1.7, platelet count <100 x 103 uL, and history or presence of ascites or hepatic encephalopathy.

* Child-bearing age women without the willing to contraceptive control, or lactating or pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver histological response | Histological response between baseline and after 144-week TAF Treatment
  Histological response is defined as an improvement of at least two points in the HAI inflammation score of Knodell necro-inflammation scoring system with no worsening of fibrosis or an improvement of at least one point in the fibrosis score of Metavir scoring system.

SECONDARY OUTCOMES:
Virology response | Virological response of 1, 2, 3 years of TAF treatment
  Virological response is defined as the percentage of patients achieve HBV DNA lower than lower detection limit.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will be shared after study completion